CLINICAL TRIAL: NCT04647084
Title: Pilot Randomized Control Trial: Comparing the Effectiveness of Buzzy Versus Intradermal Lidocaine for Peripheral Intravenous Cannulation in Adults
Brief Title: Pilot Trial: Comparing Buzzy to Intradermal Lidocaine for Peripheral IV Cannulation in Adults
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The investigators were unable to begin work on this study.
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00808
Record Dates: First submitted 2020-11-17; First posted 2020-11-30 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2022-10

CONDITIONS: Pain, Acute; Patient Satisfaction
MeSH Terms: conditions — Acute Pain; Patient Satisfaction | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intradermal Lidocaine 2% (Experimental)
  Interventions: Drug: Lidocaine 2% Injectable Solution
- Buzzy (Experimental)
  Interventions: Device: Buzzy

INTERVENTIONS:
Drug: Lidocaine 2% Injectable Solution — An elastic band will be placed around the subject's arm, and the elastic band will be removed once the IV is inserted. After the elastic band is placed on the subject's arm, the arm will be cleaned, and then a small skin wheel will be created with the lidocaine that will be injected very close to where the IV will be placed. The IV will be placed within about a minute from the time when the lidocaine was injected.
  Arms: Intradermal Lidocaine 2%
Device: Buzzy — The Buzzy vibrating ice pack will be placed on the subject's arm with an elastic band around it, and it will remain there as the arm is cleaned and prepped and the IV inserted. The Buzzy device will be removed once the IV is inserted.
  Arms: Buzzy

SUMMARY:
IV placement is necessary for surgical procedures. Unfortunately, some patients say that placing an IV is painful. The investigators are conducting this study to evaluate two techniques that could make the placement of the IV more comfortable.

DETAILED DESCRIPTION:
Currently, some medical providers administer the IV without any pain-relieving techniques. Some medical providers inject a numbing medication underneath the skin prior to the IV placement. This requires an additional needle stick. Some medical providers place a device called Buzzy® on a patient's arm prior to the IV placement. The Buzzy® device is the combination of an ice pack and a vibrator in the shape of a bumble bee. Literature shows that the Buzzy® device makes IV placement more comfortable for children, but there is minimal data in regard to whether it is helpful for adult patients.

The investigators are conducting this study to compare the effectiveness of the Buzzy® device with that of the injection of numbing medication underneath the skin for IV placement in adults. This device has been FDA approved for use.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18 to 99
2. Non-pregnant women and men
3. Adults that are able to consent
4. Patients requiring intravenous catheter insertion for their operation/procedure

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Pain with IV Cannulation based on the Visual Analog Scale | 5-20 minutes
  How much pain do adult patients experience with peripheral IV cannulation when Buzzy® device is used versus when intradermal lidocaine 2% is used? The Visual Analog Scale is used for linear measurement of pain, where the minimum number is 0 (no pain) and the maximum number is 10 (unimaginable pain).

SECONDARY OUTCOMES:
Satisfaction with IV cannulation based on the Numerical Rating Scale | 5-20 minutes
  How much satisfaction do adult patients experience with peripheral IV cannulation when Buzzy® device is used versus when intradermal lidocaine 2% is used? The Numerical Rating Scale is used for linear measurement of satisfaction, where the minimum number is 1 (very dissatisfied) and the maximum number is 5 (very satisfied).
Number of IV cannulation attempts | 5-20 minutes
  How does first attempt during peripheral intravenous cannulation in adult patients compare when Buzzy® device is used versus when intradermal lidocaine 2% is used?
Pain related to IV size based on the Visual Analog Scale | 5-20 minutes
  Does size of the peripheral intravenous catheter affect the pain that adult patients experience with peripheral IV cannulation? The Visual Analog Scale is used for linear measurement of pain, where the minimum number is 0 (no pain) and the maximum number is 10 (unimaginable pain).
Pain related to IV location based on the Visual Analog Scale | 5-20 minutes
  Does location of the peripheral intravenous catheter placement affect the pain that adult patients experience with peripheral IV cannulation? The Visual Analog Scale is used for linear measurement of pain, where the minimum number is 0 (no pain) and the maximum number is 10 (unimaginable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schoor, MD, Principal Investigator — physician
Locations (1):
- St. Elizabeth's Medical Center, Brighton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT04647084/Prot_SAP_002.pdf
  • Informed Consent Form (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT04647084/ICF_000.pdf